CLINICAL TRIAL: NCT02711917
Title: Consumption of Rocuronium Under Etomidate-based Versus Propofol-based Maintenance of General Anesthesia Under Different Concentration of Sevoflurane- BIS Guided Clinical Trial in a Closed Loop Infusion System
Brief Title: Rocuronium Consumption in Etomidate-based and Propofol-based General Anesthesia Under Sevoflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TianjinMUGH; Narina Goulvaden (Other: Tianjin medical university)
Record Dates: First submitted 2016-02-24; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Neuromuscular Monitoring
Keywords: Propofol; Sevoflurane; Etomidate; Rocuronium; BIS; Closed loop infusion system
MeSH Terms: interventions — Propofol; Etomidate; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- SP1- sevoflurane MAC 0.5 (Experimental): In this group, patient of age 40-60 years of age, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, Sevoflurane is started to achieve the desired MAC of 0.5. Propofol infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 0.5; Drug: Propofol; Drug: Rocuronium
- SP2- Sevoflurane MAC 0.75 (Experimental): In this group, patient of age 40-60 years, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen.Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, Sevoflurane is started to achieve the desired MAC of 0.75. Propofol infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 0.75; Drug: Propofol; Drug: Rocuronium
- SP3 -Sevoflurane MAC 1.0 (Experimental): In this group, patient of age 40-60 years, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, Sevoflurane is started to achieve the desired MAC of 1.0. Propofol infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 1.0; Drug: Propofol; Drug: Rocuronium
- SP4- Sevoflurane MAC 0.5 (Experimental): In this group, patient above 60 years of age, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, sevoflurane is started to achieve the desired MAC of 0.5. Propofol infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 0.5; Drug: Propofol; Drug: Rocuronium
- SP5- Sevoflurane MAC 0.75 (Experimental): In this group, patient above 60 years of age, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, Sevoflurane is started to achieve the desired MAC of 0.75. Propofol infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 0.75; Drug: Propofol; Drug: Rocuronium
- SE1- Sevoflurane MAC 0.5 (Experimental): In this group, patient of age 40-60 years of age, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, sevoflurane is started to achieve the desired MAC of 0.5. Etomidate infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 0.5; Drug: Etomidate; Drug: Rocuronium
- SE2- Sevoflurane 0.75 (Experimental): In this group, patient of age 40-60 years of age, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, sevoflurane is started to achieve the desired MAC of 0.5. Etomidate infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 0.75; Drug: Etomidate; Drug: Rocuronium
- SE3- Sevoflurane MAC 1.0 (Experimental): In this group, patient of age 40-60 years of age, ASA I/II, undergoing elective abdominal or gynecological surgery are chosen. Neuromuscular function prior to induction is assessed by acceleromyography by stimulation of ulnar nerve and noting the response of adductor pollicis. After induction and intubation, Sevoflurane is started to achieve the desired MAC of 0.5. Etomidate infusion is started to keep BIS between 40-60.
  Interventions: Drug: MAC 1.0; Drug: Etomidate; Drug: Rocuronium

INTERVENTIONS:
Drug: MAC 0.5 — 0.5 MAC Sevoflurane
  Arms: SE1- Sevoflurane MAC 0.5; SP1- sevoflurane MAC 0.5; SP4- Sevoflurane MAC 0.5
Drug: MAC 0.75 — 0.75 MAC Sevoflurane
  Arms: SE2- Sevoflurane 0.75; SP2- Sevoflurane MAC 0.75; SP5- Sevoflurane MAC 0.75
Drug: MAC 1.0 — 1.0 MAC Sevoflurane
  Arms: SE3- Sevoflurane MAC 1.0; SP3 -Sevoflurane MAC 1.0
Drug: Propofol — Propofol consumption
  Arms: SP1- sevoflurane MAC 0.5; SP2- Sevoflurane MAC 0.75; SP3 -Sevoflurane MAC 1.0; SP4- Sevoflurane MAC 0.5; SP5- Sevoflurane MAC 0.75
Drug: Etomidate — Etomidate consumption
  Arms: SE1- Sevoflurane MAC 0.5; SE2- Sevoflurane 0.75; SE3- Sevoflurane MAC 1.0
Drug: Rocuronium — Consumption of Rocuronium

SUMMARY:
Different concentration of sevoflurane was given to maintain anesthesia. The dose of propofol to maintain BIS between 40-60 and the consumption of rocuronium was recorded and evaluated.

DETAILED DESCRIPTION:
2 age group of patients was selected, 40-60 years and above 60 years. Maintenance of anesthesia was carried out using different concentration of Sevoflurane, ie MAC 0.5, 0.75 and 1.0. Bis value was kept between 40-60 and the dose of propofol required was recorded. Rocuronium infusion given in a close loop infusion system for different group was tabulated. The results was then analysed.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30
* elective Gynaecological/abdominal/urological surgery
* Operation time < 3hrs
* ASA I/II
* Intubated patients

Exclusion Criteria:

* Coronary artery disease, cardiac, lung, hepatic and renal insufficiency
* Severe uncontrolled HBP
* Obesity (BMI >30)
* Neuromuscular and metabolic diseases
* Receiving medication known to influence neuromuscular transmission
* Pregnancy
* Psychiatric disorders
* Allergy history to any of the drugs that will be used

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
consumption of propofol | Intraoperative
  Propofol, Etomidate, Rocuronium consumption under specific concentration of sevoflurane keeping BIS between 40-60

SECONDARY OUTCOMES:
Recovery Index | Intraoperative
  T25%-T75%
Onset time | Intraoperative
  Time from starting infusion of Rocuronium at induction till T<10%
Sevoflurane time | Intraoperative
  Time from starting sevoflurane till end tidal concentration is reached

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, Professor, Principal Investigator — Head of department anesthesiology

IPD SHARING:
Plan to Share IPD: Undecided